CLINICAL TRIAL: NCT03484650
Title: Systemic Lidocaine Infusion for Pain Control in Ventral Hernia
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of available resources to complete study
Sponsor: Carilion Clinic (Other)
Responsible Party: Principal Investigator, Curtis Bower, Vice Chief of Carilion Clinic General Surgery, Carilion Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2344
Record Dates: First submitted 2018-03-26; First posted 2018-04-02 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The patient, physician, and data abstractors will be blinded to the arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Placebo Comparator): Patients will receive standard care plus infusion of placebo
  Interventions: Other: Placebo
- Lidocaine (Experimental): Patients will receive lidocaine infusions peri-operatively
  Interventions: Drug: Lidocaine Hydrochloride

INTERVENTIONS:
Drug: Lidocaine Hydrochloride — Lidocaine bolus to be given 1 hour pre-operatively
  Other Names: Bolus of lidocaine
  Arms: Lidocaine
Drug: Lidocaine Hydrochloride — Lidocaine infusion will be started after the bolus and be continued for 24 hours post-operatively
  Other Names: Infusion of lidocaine
  Arms: Lidocaine
Other: Placebo — Control patients will receive a placebo bolus and infusion of saline to match the experimental arm.
  Arms: Control

SUMMARY:
Ventral hernia repair leads to more than expected pain. This is thought to be secondary to nerve pain at the lateral transfixion sutures. Systemic lidocaine given pre-op has in other situations decreased neurogenic pain. This study will examine its effects on pain experienced after ventral hernia repair.

DETAILED DESCRIPTION:
Patients presenting to the surgical clinic for elective repair of ventral hernia defects will be offered the opportunity to participate in a study that aims to reduce post-operative pain. Benefits and risks will be discussed with the patient, and the patient will understand that their decision to opt in or opt out will not affect the minimum standard of care. Once agreeable, the patient will undergo pre-infusion assessment. Such pre-operative evaluation will include complete pain history, quantitative pain assessment, medical history, physical exam, electrocardiogram, and laboratory workup. Specific workup will focus on heart failure or liver disease, as these increase the toxicity of lidocaine. Nevertheless, the low dose of infusion planned is not contraindicated with heart or liver disease. Patients will then be assigned equally and randomly to experimental and control groups. Physicians will be blinded from these assignments. The experimental patient will be treated with IV lidocaine bolus of 1.5 mg/kg and thereafter with infusion at 0.5 mg/kg/hour. Infusion will begin at least one hour prior to incision and continued for 24 hours after incision, unless adverse reactions experienced. Post-operative pain in eight-hour increments will be recorded. Additional opiates required to control pain during admission and after discharge will be recorded. Length of hospital stay will also be documented. The electronic medical record will be utilized to collect the below parameters. The control group will receive standard of care, along with placebo volume and rate of administration of saline equivalent to the volume and rate of the lidocaine infusion. To monitor inpatient pain medication, each patient in the control and experimental group will be prescribed the same analgesia PRN orders. The MAR feature in the electronic patient record will allow determination of the amount of PRN pain medication doses required by each patient. Physicians will be blinded and continue to adjust pain medication orders as needed for optimal patient care. Narcotic requirements for each patient can be standardized to morphine equivalents for analysis.

To monitor outpatient pain medication, each patient in the control and experiential group upon discharge will be given the same analgesia prescriptions, e.g. oxy 5 mg dips #30. Patients will bring back their bottles of pills to be counted at the 2-week post-operative visit. The investigators will call patients at the 30th post-operative day to see how much of the pain medication is in continued use.

ELIGIBILITY:
Inclusion Criteria:

Age over 18 Ventral hernia Elective operation Surgeon anticipates mesh

-

Exclusion Criteria:

Age less than 18 Incapable of informed consent Comorbid condition that precludes lidocaine Pregnancy Emergency procedures No mesh History of narcotic abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain | 30 days
  Amount of morphine equivalents opioid medication used 30 days post-op

CONTACTS AND LOCATIONS:
Overall Officials: Sandy L Fogel, MD, Principal Investigator — Carilion Clinic
Locations (1):
- Carilion Roanoke Memorial Hospital, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
No data to be shared.